CLINICAL TRIAL: NCT05990764
Title: Effects of a Combination of Polyphenol-rich Extracts, Prebiotics, and Hydrolyzed Fiber on the Quality of Life of Patients With Irritable Bowel Syndrome (IBS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AronPharma Sp. z o. o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 03-AP-IBS
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: IBS; Gastrointestinal diseases; Probiotic; Prebiotic; Plant extract; Polyphenol-rich Extracts
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases | interventions — Probiotics; Prebiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Probiotic, Prebiotic, Polyphenol-rich Extracts (Experimental): 18 patients with IBS
  Interventions: Dietary Supplement: Probiotic, Prebiotic, Polyphenol-rich Extracts
- Probiotic, Prebiotic (Experimental): 18 patients with IBS
  Interventions: Dietary Supplement: Probiotic, Prebiotic
- Placebo (Placebo Comparator): 18 patients with IBS
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic, Prebiotic, Polyphenol-rich Extracts — probiotic strains, prebiotic (Partially Hydrolyzed Guar Gum) and elderberry and chokeberry extract
  Once a day
  Arms: Probiotic, Prebiotic, Polyphenol-rich Extracts
Dietary Supplement: Probiotic, Prebiotic — probiotic strains, prebiotic (Partially Hydrolyzed Guar Gum)
  Once a day
  Arms: Probiotic, Prebiotic
Other: Placebo — placebo
  Once a day
  Arms: Placebo

SUMMARY:
The aim of the study is to demonstrate a beneficial effect in reducing symptoms that negatively affect the quality of life of IBS patients, and to demonstrate a positive effect on inflammatory and intestinal function markers.

DETAILED DESCRIPTION:
The double-blind, randomized, placebo-controlled study will be conducted on 48 patients (18-55 years old) with Irritable Bowel Syndrome (IBS). The study will consist of 2 months of supplementation with three parallel arms: 1) probiotic strains and prebiotic (Partially Hydrolyzed Guar Gum); 2) probiotic strains, prebiotic (Partially Hydrolyzed Guar Gum) and elderberry and chokeberry fruit extract; 3) placebo.The study will assess symptoms associated with IBS, using the IBS-QOL questionnaire and the Bristol Stool Formation Scale. Markers of inflammation and intestinal barrier permeability , will be determined in blood and stool samples collected from patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Irritable Bowel Syndrome.
* Women and men, 18-55 years old.
* Signed informed consent.

Exclusion Criteria:

* Intake of supplements containing plant extracts, polyphenols or anthocyanins, and supplements containing fiber, probiotics and prebiotics.
* Participation in another clinical trial.
* Inability to swallow an oral study drug/placebo.
* Oncological disease, autoimmune disease, severe liver dysfunction, tuberculosis, leukemia, multiple sclerosis, AIDS, rheumatoid arthritis, organ transplant and other gastrointestinal diseases that may affect the results of the study.
* Women who are pregnant, planning to become pregnant during the study, or breastfeeding,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
IBS-QoL (Irritable Bowel Syndrome-Quality of Life) index | Baseline, 2 months
  IBS-QoL measures the impact of the disease on the quality of life of patients with IBS
Stool consistency | Baseline, 2 months
  Will be assessed using the Bristol Stool Chart

SECONDARY OUTCOMES:
Zonulin | Baseline, 2 months
  Zonulin level in stool samples
Short-chain fatty acids | Baseline, 2 months
  Short-chain fatty acids level in stool samples
IL-6 | Baseline, 2 months
  IL-6 level in serum samples
IL-8 | Baseline, 2 months
  IL-8 level in serum samples
I-FABP | Baseline, 2 months
  I-FABP level in serum samples

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No